CLINICAL TRIAL: NCT00773552
Title: Randomized Double Blinded Placebo-controlled Trial of the Once Daily 5mg Dose of Solifenacin Succinate vs. Placebo in Inner City Women Ages 20-45 With Overactive Bladder
Brief Title: Solifenacin Succinate Versus Placebo in Inner City Women Ages 20-45 With Overactive Bladder
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator Left Institution
Sponsor: Stamford Hospital (Other)
Responsible Party: Anthony Gaddi M.D., The Stamford Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-0917.01
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Urinary Urge; Urge Incontinence; Overactive Bladder
Keywords: OAB; overactive bladder; urinary urge; urge incontinence; urge
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Bladder, Overactive | interventions — Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- solifenacin succinate (Experimental): Group randomized into solifenacin succinate treatment
  Interventions: Drug: solifenacin succinate
- placebo (Placebo Comparator): Group randomized into placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: solifenacin succinate — 5mg PO Qday x 90 days
  Other Names: VESIcare
  Arms: solifenacin succinate
Drug: placebo — 1 tab PO Qday x 90 days
  Arms: placebo

SUMMARY:
In this study we hope to establish the prevalence of urinary urge symptoms (with or without incontinence) in a multicultural, underserved, hospital clinic population in women between the ages of 20 and 45. Quality of life (QOL) in these individuals will be examined. The goal is to show a 15% reduction in number of voids in a 24 hour period in our study population after 12 weeks of treatment with solifenacin succinate.

Hypothesis: We believe that urinary urge symptoms are under-reported in young women and believe they pose a significant strain on quality of life on otherwise young, healthy individuals. Treatment with solifenacin succinate will improve symptoms, in turn improving QOL for these individuals.

DETAILED DESCRIPTION:
* Study type: 1) Prospective, questionnaire based study 2) Randomized, double blinded, placebo-controlled trial
* Setting: OB-GYN, general medicine, and family medicine clinics at the Stamford Optimus Health Clinic in association with The Stamford Hospital Department of OB-GYN.
* Study population: Pre-menopausal women, ages 20-45
* Number of patients: 40 in each treatment arm (n=80)
* Recruitment: Questionnaire based, handed out by our research assistant to any women visiting Optimus Health Clinics (general medicine, family medicine, and OB-GYN) regardless of reason for visit. Follow up visits for qualifying individuals will be held in the department of OB-GYN at The Stamford Hospital.

Subject Compensation: Subjects will receive $10 for filling out the initial questionnaires. If the subject proceeds to the treatment arm of the study, they will be given $50 a month (total of $150) during the 90 day treatment period.

* Study Treatment: Placebo-controlled medical treatment with solifenacin succinate, 5mg PO Qday x 90 days.
* Randomization/blinding method/drug administration: The Stamford Hospital pharmacy will be in charge of blinding treatment to both researchers and study population. The drug and placebo will both be stored and administered by the pharmacy. A computer randomization software will be used by the pharmacy to randomize patients. The subjects will be dispensed a one month supply of drug/placebo at a time. The subsequent months refill will be administered only if the patient brings the original container back to the pharmacy so that compliance can be tracked. Both placebo and solifenacin succinate will be supplied by Astellas Pharmaceuticals and will look identical.
* Primary endpoint: subjects will remain in study up to 120 days (90 days of treatment, and up to 30 days allotted for scheduling initial visit, history and physical, obtaining consent, etc).
* Primary Goal: 15% reduction in the number of voids in a 24 hour period after 12 weeks of treatment with Solifenacin succinate.
* Secondary Goals:
* Determining prevalence of urinary urge symptoms in pre-menopausal women ages 20-45.
* Assessing quality of life prior to treatment with respect to urge symptoms, then monitoring for improvement after treatment.
* Decreases in the relative number of episodes of: urgency, nocturia (defined as waking 1 or more times to urinate per night14), and incontinence.
* Reported (using 3-day diary) medical side effects including: complaints of dry mouth, constipation, and blurred vision.

Statistical Considerations:

With the above stated worldwide urinary urge symptom prevalence found to be 16-17%, we are attempting to show a reduction of 15% in urinary urge symptoms, using an alpha of 0.05 with a power of 80%. Calculated sample size was determined to be 68, 34 in the medical arm and 34 in the placebo arm. The overall goal for enrollment will be increased to 80 to account for possible study drop outs.

Methods:

This study will be a 3 tiered, prospective study looking at urinary urge symptoms (with and without incontinence). Pre-menopausal women between the ages of 20-45, will be given a validated urge incontinence questionnaire (OAB-V82 ) at time of visit to the Optimus OB-GYN, General Medicine, and Family Medicine clinics, regardless of reason for visit.

Patients with a score of 8 or greater on the OAB-V8 will be selected out for inclusion into our study. Exclusions for this study are as mentioned above. Patients on anticholinergics/antimuscarinics will undergo a 2 week washout period prior to inclusion into treatment arms. From this data, prevalence of urinary urge symptoms will be calculated.

The study group will then be given another validated questionnaire (King's Health Questionnaire3, 5 or KHQ) to analyze quality of life given their urge symptoms prior to randomization. This will be quantified using the scoring system associated with the KHQ. The above mentioned questionnaires will be written in three of the most common languages in our population including English, Spanish, and French. If translation is necessary, the language line will be used. Translator number and name will be obtained for records.

A pregnancy test will be administered prior to treatment, which will be supplied by the department of OB-GYN (if the subject were to become pregnant during the study, the patient is to contact one of the study investigators immediately since it is a class C drug). We will then randomize subjects into one of two treatment arms, medical or placebo; using the antimuscarinic drug solifenacin succinate 5mg po Qday for a 12 week period. The Stamford Hospital pharmacy will be in charge of blinding, randomization, storage of drug and placebo, and administration of medication (as described above).

This dosage has not only been shown to significantly improve urinary urge symptoms, but it is also well tolerated and has a more favorable side effect profile3,12. In general, solifenacin succinate has been shown to be efficacious in reducing overactive bladder related symptoms3, 7-10, 12, 13.

The treatment outcomes will then be compared to examine improvement in symptoms. Subjects will have an initial visit (for obtaining consent, brief history and physical, explaining study, etc.), then monthly follow up visits once treatment is initiated. These visits will be held in the department of OB-GYN in The Whittingham Pavillion at The Stamford Hospital. A 3 day urinary diary will be filled out at the end of each month of treatment and brought to follow up visits in order to quantify improvement/reduction in urinary urge symptoms. We will also re-evaluate patients upon completion of treatment for improvement of QOL and urge symptoms using the KHQ.

ELIGIBILITY:
Inclusion Criteria:

* Score of 8 or greater on the OAB-V8 questionnaire
* Women between the ages of 20 and 45 years.
* Pre-menopausal
* Not Pregnant or plan on becoming during the length of the study

Exclusion Criteria:

* menopause
* pregnancy (including women breastfeeding, or women planning on becoming pregnant during the study); a pregnancy test will be performed prior to starting treatment.
* previous diagnosis of stress urinary incontinence or mixed urinary incontinence
* previous diagnosis of diabetes mellitus/diabetes insipidus
* use of diuretics
* neurological cause for detrusor instability
* medical condition contraindicating antimuscarinic use (i.e.: narrow angle glaucoma)
* urinary tract infection/cystitis/bladder stones (at time of questionnaire).
* taking any of the following contraindicated drugs:

  1. cisapride
  2. phenothiazines: fluphenazine or fluphenazine decanoate, prochlorperazine maleate, promethazine, chlorpromazine, perphenazine, thioridazine, trifluoperazine, prochlorperazine edisylate,
  3. pimozide
  4. potassium salts: potassium acid phosphate, potassium citrate, potassium chloride, potassium iodide, potassium phosphate/sodium potassium.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
15% reduction in the amount of voids in a 24 hour period | 90 days

SECONDARY OUTCOMES:
Assessing quality of life prior to treatment with respect to urge symptoms, then monitoring for improvement after treatment. | 90 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Optimus Health care, Stamford, Connecticut
  - The Stamford Hospital, Stamford, Connecticut